CLINICAL TRIAL: NCT02675257
Title: Depression and Diabetes Control Trial
Acronym: DDCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Collaborators: German Center for Diabetes Research (Other); Helmholtz Zentrum München (Industry); German Diabetes Center (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Norbert Hermanns, Prof. Dr. phil. Norbert Hermanns, Forschungsinstitut der Diabetes Akademie Mergentheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FKZ 82DZD01101
Record Dates: First submitted 2016-02-02; First posted 2016-02-05 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus; Affective Disorders; Depression; Depressive Symptoms; Emotional Distress; Diabetes Complications
Keywords: Diabetes mellitus; Affective disorders; Depressive symptoms; Diabetes distress; Hyperglycaemia; Dysglycaemia; Glycaemic control; Self-care behaviour; Quality of Life; Diabetes acceptance; Diabetes complications; Low-grade inflammation; Inflammatory markers; Stress reactivity; Health-care costs
MeSH Terms: conditions — Diabetes Mellitus; Mood Disorders; Depression; Diabetes Complications; Hyperglycemia | interventions — Delivery of Health Care; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive-behavioural group treatment (Experimental): Five group sessions of diabetes-Specific cognitive-behavioural group treatment for diabetes patients with depressive symptoms and/or diabetes distress and suboptimal glycaemic control.
  Interventions:
  * Diabetes-related affective problems analysis
  * Goal setting towards improvement of glycaemic control
  * Diabetes-specific problem-solving therapy
  * Interventions to increase diabetes treatment motivation
  * Activation of personal and social resources
  * Reduction of barriers to self-care/glycaemic control
  * Cognitive restructuring of diabetes-related problems
  * Goal definition regarding self-care/glycaemia/well-being
  Interventions: Behavioral: Diabetes-related affective problems analysis; Behavioral: Goal setting towards improvement of glycaemic control; Behavioral: Diabetes-specific problem-solving therapy; Behavioral: Interventions to increase diabetes treatment motivation; Behavioral: Activation of personal and social resources; Behavioral: Reduction of barriers to self-care/glycaemic control; Behavioral: Cognitive restructuring of diabetes-related problems; Behavioral: Goal definition regarding self-care/glycaemia/well-being
- Treatment-as-usual (Active Comparator): Standard diabetes education.
  Interventions:
  * Health care and specific topics (e. g. blood pressure)
  * Healthy foods, cooking recommendations, recipes
  * Sports, activities and exercise
  * Foot care: exercises, care & control, injuries, neuropathy
  * Diabetes complications
  * Social aspects of living with diabetes
  Interventions: Behavioral: Health care and specific topics (e. g. blood pressure); Behavioral: Healthy foods, cooking recommendations, recipes; Behavioral: Sports, activities and exercise; Behavioral: Foot care: exercises, care & control, injuries, neuropathy; Behavioral: Diabetes complications; Behavioral: Social aspects of living with diabetes

INTERVENTIONS:
Behavioral: Diabetes-related affective problems analysis — Analysis of diabetes-related affective problems with regard to suboptimal glycaemic control
  Arms: Cognitive-behavioural group treatment
Behavioral: Goal setting towards improvement of glycaemic control — Discussing and setting goals regarding improvements of suboptimal glycaemic control, depressive symptoms and diabetes distress
  Arms: Cognitive-behavioural group treatment
Behavioral: Diabetes-specific problem-solving therapy — Diabetes-specific problem-solving therapy with main focus on suboptimal glycaemic control, depressive symptoms and diabetes distress
  Arms: Cognitive-behavioural group treatment
Behavioral: Interventions to increase diabetes treatment motivation — Interventions to increase diabetes treatment motivation in order to achieve improvements of glycaemic control as well as recovery from affective problems
  Arms: Cognitive-behavioural group treatment
Behavioral: Activation of personal and social resources — Activation of personal and social resources with a view to diabetes control and affective problems
  Arms: Cognitive-behavioural group treatment
Behavioral: Reduction of barriers to self-care/glycaemic control — Definition and reduction of barriers to adequate diabetes self-care behaviour as well as good glycaemic control
  Arms: Cognitive-behavioural group treatment
Behavioral: Cognitive restructuring of diabetes-related problems — Cognitive restructuring of diabetes-related problems such as suboptimal glycaemic control and diabetes-related affective problems
  Arms: Cognitive-behavioural group treatment
Behavioral: Goal definition regarding self-care/glycaemia/well-being — Goal definition and agreement regarding diabetes self-care behaviour, optimal glycaemic control and activities supporting well-being and recovery from affective symptoms
  Arms: Cognitive-behavioural group treatment
Behavioral: Health care and specific topics (e. g. blood pressure) — Education on health care and specific topics (e. g. blood pressure)
  Arms: Treatment-as-usual
Behavioral: Healthy foods, cooking recommendations, recipes — Education on healthy and unhealthy foods, cooking and recipes
  Arms: Treatment-as-usual
Behavioral: Sports, activities and exercise — Education on sports, activities and exercise
  Arms: Treatment-as-usual
Behavioral: Foot care: exercises, care & control, injuries, neuropathy — Education on foot care: exercises, care and control, injuries, and diabetic neuropathy
  Arms: Treatment-as-usual
Behavioral: Diabetes complications — Education on diabetes complications
  Arms: Treatment-as-usual
Behavioral: Social aspects of living with diabetes — Education on social aspects of living with diabetes
  Arms: Treatment-as-usual

SUMMARY:
This randomised controlled trial evaluates a cognitive-behavioural intervention for diabetes patients with suboptimal glycaemic control and comorbid depressive symptoms and/or diabetes distress. The main outcome is the improvement of suboptimal glycaemic control (HbA1c). Secondary outcomes are effects on depressive symptoms, diabetes distress, self-care behaviour, diabetes acceptance and quality of life. The treatment group will be treated with a cognitive-behavioural group treatment comprising specific interventions to improve glycaemic control and reduce diabetes distress as well as depressive symptoms. The control group will receive treatment-as-usual. A total of 212 study participants will be included. A secondary study objective is to analyse associations of suboptimal glycaemic control, depressive symptoms and diabetes distress with inflammatory markers.

DETAILED DESCRIPTION:
Suboptimal glycaemic control is an established risk factor for the development of serious long-term complications of diabetes. Moreover, it is associated with elevated risks of significant hyperglycaemic acute events such as hyperosmolar hyperglycemic state or diabetic ketoacidosis. Hence, patients with diabetes and persistent suboptimal glycaemic control are at higher risk of having a rather poor prognosis.

Besides physiological and medical factors, psychological problems have been found to predict suboptimal glycaemic control. A number of studies found depressive symptoms to be independently associated with hyperglycaemia. Others focussed on diabetes-specific affective problems - the so called diabetes distress - and suggested this factor to be of great importance. Finally, some studies found that depressive symptoms and diabetes distress may interact, with the coocurrence of these factors being associated with the highest risk or suboptimal glycaemic control. The results correspond to other findings suggesting that both depressive symptoms and diabetes distress are often associated with reduced diabetes self-care, which can explain the associations of those factors with hyperglycaemia.

On the other hand, suboptimal glycaemic control could also be an explanation for affective problems - either mediated by physiological mechanisms or psychological ones, e.g. dissatisfaction or guilt. Hence, it is valid to assume that the link between depressive symptoms and/or diabetes distress may be bidirectional - although evidence to support this assumption is missing.

Following this evidence and background, the investigators designed the a to analyse the relationships between suboptimal glycaemic control, depressive symptoms and diabetes distress in diabetes using a prospective study design. The study is a randomized trial in which a cognitive-behavioural group treatment is compared to a treatment-as-usual condition (standard diabetes education) regarding their efficacy in improving suboptimal glycaemic control. 212 diabetes patients with suboptimal glycaemic control (HbA1c value > 7.5%) and elevated depressive symptoms (Center for Epidemiologic Studies Depressions Scale score ≥ 16) and/or elevated diabetes distress (Problem Areas In Diabetes Scale score ≥ 40) will be randomly assigned to either the treatment group or treatment-as-usual. The primary outcome is the improvement of suboptimal glycaemic control (reduction of HbA1c) in the 12-month follow-up. As secondary outcomes positive baseline-to-follow up changes regarding depressive symptoms, diabetes distress, diabetes self-care behaviour, diabetes acceptance and quality of life are assessed.

A second study objective is to analyse cross-sectional and prospective associations of suboptimal glycaemic control, depressive symptoms and diabetes distress with serum levels of the following inflammatory markers: hsCRP, IL-6, IL-18, IL-1Ra, MCP-1 and Adiponectin. Potential effects of the treatment groups on these markers will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70
* Diabetes mellitus type 1 or type 2
* Diabetes duration ≥ 1 year
* Suboptimal glycaemic control (HbA1c > 7,5%)
* Elevated depressive symptoms (CES-D score ≥ 16) and/or elevated diabetes distress (PAID score ≥ 40)
* Sufficient language skills
* Written informed consent

Exclusion Criteria:

* Severe major depressive disorder according to ICD-10
* Current psychiatric and/or psychotherapeutic treatment
* Current antidepressive medical treatment
* Suicidal ideation
* Acute mental disorder of the following type: schizophrenia or other psychotic disorder, bipolar disorder, severe eating disorder (anorexia nervosa, bulimia nervosa), substance use disorder
* History of personality disorder
* Severe somatic illnesses: dialysis-dependent nephropathy, acute cancer, severe heart disease (NYHA III - IV), severe neurologic illness (e. g. MS, dementia), severe autoimmune disease
* Terminal illness
* Bedriddenness
* Guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Improvement of glycaemic control as measured by the HbA1c | 12 months
  Mean difference between HbA1c values at baseline and at 12 month follow

SECONDARY OUTCOMES:
Improvement of glycaemic control as measured by participants' blood glucose meter or glucose monitoring devices (data are extracted from tools using the diasend application) | 12 months
  Mean difference between average glucose test scores during an 8-week period before baseline and those during an 8-week period before 12 month follow
Improvement of depressive symptoms as measured with the Center for Epidemiologic Studies Depression Scale (CES-D) | 12 months
  Mean difference between CES-D scores at baseline and at 12 month follow up
Improvement of depressive symptoms as measured with the Patient Health Questionnaire Module for Depression (PHQ-9) | 12 months
  Mean difference between PHQ-9 scores at baseline and at 12 month follow up
IImprovement of diabetes distress as measured with the Problem Areas in Diabetes Scale (PAID) | 12 months
  Mean difference between PAID scores at baseline and at 12 month follow
IImprovement of diabetes distress as measured with the Diabetes Distress Scale (DDS) | 12 months
  Mean difference between DDS scores at baseline and at 12 month follow
Improvement of self-care behaviour as measured with the Summary of Diabetes Self-Care Activities Measure (SDSCA) | 12 months
  Mean difference between SDSCA scores at baseline and at 12 month follow
Improvement of self-care behaviour as measured with the Diabetes Self-Management Questionnaire (DSMQ) | 12 months
  Mean difference between DSMQ scores at baseline and at 12 month follow
Improvement of diabetes acceptance as measured with the Diabetes Acceptance Scale (DAS) | 12 months
  Mean difference between DAS scores at baseline and at 12 month follow
Improvement of quality of life as measured with the EuroQol Five-Dimensions Questionnaire (EQ-5D) | 12 months
  Mean difference between EQ-5D scores at baseline and at 12 month follow
Improvement of quality of life as measured with the Short Form-36 Health Survey (SF-36) | 12 months
  Mean difference between SF-36 scores at baseline and at 12 month follow

OTHER OUTCOMES:
Inflammatory Marker: hsCRP | 12 months
  Mean difference between hsCRP scores at baseline and at 12 month follow
Inflammatory Marker: IL-6 | 12 months
  Mean difference between IL-6 scores at baseline and at 12 month follow
Inflammatory Marker: IL-18 | 12 months
  Mean difference between IL-18 scores at baseline and at 12 month follow
Inflammatory Marker: IL-1Ra | 12 months
  Mean difference between IL-1Ra scores at baseline and at 12 month follow
Inflammatory Marker: MCP-1 | 12 months
  Mean difference between MCP-1 scores at baseline and at 12 month follow
Inflammatory Marker: Adiponectin | 12 months
  Mean difference between Adiponectin scores at baseline and at 12 month follow

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Haak, Prof., MD, Principal Investigator — Diabetes Center Mergentheim
Locations (2):
- Germany (2):
  - Diabetes Center Mergentheim, Bad Mergentheim, Baden-Wurttemberg
  - Forschungsinstitut der Diabetes Akademie Mergentheim e. V., Bad Mergentheim, Baden-Wurttemberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmitt A, Ehrmann D, Kuniss N, Muller N, Kulzer B, Hermanns N. Assessing fear of complications in people with type 1 and type 2 diabetes with the Fear of Diabetes Complications Questionnaire. Health Psychol. 2023 Sep;42(9):674-685. doi: 10.1037/hea0001304. Epub 2023 Jul 27. PMID 37498716